CLINICAL TRIAL: NCT01026532
Title: Functional Activity of Airway Eosinophils in Allergic Disease
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2014-1481; H-2009-0050 (Other: UW HS IRB); P01HL088594 (NIH)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Segmental antigen challenge: Segmental allergen challenge: Briefly, this procedure will be done during a bronchoscopy. Two airway tubes of the lung will have about 1 teaspoon of allergen put in it while the scope is wedged in an airway tube segment. The allergen will stimulate this portion of the airway tube to produce eosinophils. The scope will then be removed. The bronchoscopy will be repeated two days later to collect lung fluid and biopsy samples from the parts of the lung where the allergen solution was placed.
  Interventions: Biological: Segmental Allergen Challenge

INTERVENTIONS:
Biological: Segmental Allergen Challenge — Segmental allergen challenge: Briefly, this procedure will be done during a bronchoscopy. Two airway tubes of the lung will have about 1 teaspoon of allergen put in it while the scope is wedged in an airway tube segment. The allergen will stimulate this portion of the airway tube to produce eosinophils. The scope will then be removed. The bronchoscopy will be repeated two days later to collect lung fluid and biopsy samples from the parts of the lung where the allergen solution was placed.

SUMMARY:
The purpose of this study is to determine how a special white blood cell, the eosinophil, can contribute to asthma. One of the characteristics of asthma is airway inflammation. Airway inflammation in asthma may occur when an allergen is inhaled and sets up an allergic reaction in the bronchial tubes. This reaction may lead to chest tightness, cough and wheeze. To better understand the way in which the eosinophil can cause inflammation, the investigators plan to study eosinophils that move in to the lung following an allergic reaction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Diagnosis of allergic rhinitis and/or mild asthma
* Pre-albuterol forced expiratory volume in the first second (FEV1) of >70% predicted.
* Skin test positive to house dust mite (D. farinae), short ragweed or cat hair
* Documented negative Tuberculin skin test (PPD) within the last 12 months or a medical history that is consistent with a low probability of exposure to tuberculosis (i.e. the subject is not a health worker, has not traveled to endemic areas, and has no pre-existing medical or social risk factors for tuberculosis).
* At least a 20% decrease in FEV1 during the immediate response following inhaled antigen challenge
* Safety laboratory assessments within normal ranges (labs to include complete blood count with differential, blood urea nitrogen, creatinine, Prothrombin time, Partial Thromboplastin Time and platelet count)
* Women of child-bearing potential (WCBP) must have a negative urine pregnancy test (urine HCG) within 48 hours of the methacholine challenge at Visit 2, within 48 hours of the inhaled allergen challenge at V3 and on the day of the segmental allergen challenge on Visit 5. WCBP must agree to use a reliable method of birth control for the duration of the study (reliable methods of birth control can include abstinence, barrier methods, oral contraceptives, injection contraceptives or skin absorption contraceptives).
* In the opinion of the investigator, capable and willing to grant written informed consent and cooperate with study procedures and requirements

Exclusion Criteria:

* Major health problems such as autoimmune disease, heart disease, type I and II diabetes, uncontrolled hypertension or lung diseases other than asthma. The listed health problems are definitive exclusion but decisions regarding major health problems not listed will be based upon the judgment of the investigator.
* No pre-existing chronic infectious disease.
* Any condition for which, in the opinion of the investigator, transient oxyhemoglobin desaturation is inadvisable.
* Pregnant or lactating females or has a planned pregnancy during the course of the study.
* Medication other than for asthma, allergies or contraception (e.g. monoamine oxidase inhibitors and beta-adrenergic antagonists in any form).
* Inhaled corticosteroids or oral corticosteroids within 1 month of screening.
* Upper or lower respiratory infection within 1 month of screening.
* Unstable asthma as indicated by self report of increased symptoms or increased beta-agonist use over the 2 weeks preceding the screening visit.
* Current smokers (defined as smoked within the last year) or a former smoker with a history of >5 pack years.
* Obesity as defined by a Body Mass Index (BMI) >30.
* Use of an investigational drug within 30 days of entering the study
* History of noncompliance with medical regiments or subjects who are considered unreliable including those with a psychiatric history that, in the opinion of the investigator, may interfere with the conduct of study procedures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Well-controlled allergic subjects with mild-intermittent asthma will be identified and undergo inhaled allergen provocation to demonstrate an allergen-specific airway response.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-08-24 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is to use segmental antigen challenge by bronchoscopy to elicit airway eosinophilia and to retrieve cells from the airway for analysis of their function. | 48 hours
  Measurement taken at 48 hours after segmental antigen challenge.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes